CLINICAL TRIAL: NCT04651270
Title: Assessment of the Wide Field of View Provided by the SurroundScope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: 270Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL 0334
Record Dates: First submitted 2020-11-17; First posted 2020-12-03 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Laparoscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SurroundScope (Experimental): For laparoscopic camera system, the SurroundScope. 270-degree angle videoscope (270Surgical, Israel) was used
  Interventions: Device: SurroundScope

INTERVENTIONS:
Device: SurroundScope — The study will evaluate standard laparoscopic surgery using the 270Surgical system. The procedure will be performed according to the institution's standard of care, using the SurroundScope for visualization.

SUMMARY:
The aim of this study is to assess the need and potential benefits of the wide field of view during general and gynecology laparoscopic surgery.

DETAILED DESCRIPTION:
The tremendous popularity of the laparoscopic surgeries is balanced with its tradeoffs - the needs for an excellent intracavitary visualization along with a surgeon skill set capable of performing these, often more technically challenging procedures. Image quality has improved, but there are still various restrictions to images captured by the lens at the tip of a long tubular laparoscope.

270Surgical developed a 270 degree angle scope to overcome these unmet needs and improve the image quantity and extent during laparoscopy. The study will evaluate standard laparoscopic surgery using the 270Surgical system; "The SurroundScope".

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18
2. Capable of giving informed consent
3. Scheduled for general or gynecology laparoscopic surgery or open procedure that in the surgeon's opinion can be performed laparoscopically with the 270System

Exclusion Criteria:

1. Unfit for surgery: concomitant disorders incompatible with the study or surgery (at the discretion of the investigator)
2. Patients with contraindications to undergo surgery
3. Patients with ASA class* >3
4. Advanced cirrhosis with failure of hepatic function
5. Patients who have participated in another interventional clinical study in the last month
6. Pregnancy
7. Unable to consent (due to cultural, language or neurological barriers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the need and potential benefits of the wide field of view | Day of surgery
  Assessed by a multi-question subjective questionnaire completed in the OR, immediately after the case, by the surgeon and the camera person and constructed on a Likert-type, 5-point scale (1=Strongly disagree, 2=Disagree, 3=Neither agree or disagree, 4=Agree, 5=Strongly agree).

SECONDARY OUTCOMES:
Assessment of the 270 Lenses clearance contribution to the procedure. | Day of surgery
  Lenses clearance contribution will be assessed by:
  Rating of the visual impairment due to smoke using a likert-type scale of 1-5: 1=imperceptible, 2= perceptible but not interfering, 3=same as in standard procedure, 4=annoying, 5=Very annoying.
Assessment of the 270 Lenses clearance contribution to the procedure. | Day of surgery
  Lenses clearance contribution will be assessed by:
  Amount of removals and pauses for fog and smoke incidences using a scale of 1-5: 1=none, 2= less than in standard procedure, 3=same as in standard procedure, 4= more than in standard procedure, 5=much more than in standard procedure.
A record of complications related to the SurroundScope | Day of surgery up to 2 weeks after the surgical procedure
  The SurroundScope related operative complications, that require further clinical intervention

OTHER OUTCOMES:
Additional measurements - timing, compared to retrospective data of matched anonymous 100 patients' data from the medical records of the hospital. | day of surgery
  Measuring time of laparoscopic procedure (lap inserted to final lap removal)
Additional measurements- Intraoperative events | day of surgery
  Measurements include collecting a log of events that could have been missed with standard scope and were captured in the side screens
Additional measurements - lengs of stay, compared to retrospective data of matched anonymous 100 patients' data from the medical records of the hospital. | Up to two weeks
  Number of days patients stayed at the hospital following the operation

CONTACTS AND LOCATIONS:
Overall Officials: Gideon Sroka, MD, Principal Investigator — Bnai Zion Medical Center, 47 Golomb St. Haifa, 31048, Israel
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel